CLINICAL TRIAL: NCT02198859
Title: Phase 1 Study of Evaluation of Lithium and it's Effect on Clinically Localized Prostate Cancer.
Brief Title: Evaluation of Lithium and It's Effect on Clinically Localized Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13582
Record Dates: First submitted 2014-07-07; First posted 2014-07-24 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Lithium; Androgen; PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithium (Experimental): Oral lithium carbonate dose escalation: Level 1 of 600 mg/day, then escalating to Level 2 of 900 mg/day, then the final Level 3 of 1200 mg/day.
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate

SUMMARY:
Laboratory testing has suggested that lithium may decrease the incidence of certain types of cancer, including prostate cancer. Additional research has suggested that lithium decreases prostate cancer tumor size over time. This study will investigate the effect of lithium on men with prostate cancer.

DETAILED DESCRIPTION:
As lithium has been shown in an in vitro model to suppress cellular proliferation, and suppress tumor growth in an in vivo xenograft model, we propose to determine its effect on prostate cancer cells in human patients undergoing radical prostatectomy. In this pilot study we plan to assess the toxicity of lithium administration in patients prior to radical prostatectomy. This will include any clinical toxicity as well as any increase in intra-, peri- or postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent form.
* Subjects with histologically confirmed local adenocarcinoma of the prostate who have elected to proceed with radical prostatectomy as primary curative therapy.
* Subjects having no prior administration of lithium or lithium containing medications within 90 days of study enrollment.
* Subjects >/= 18 years of age.
* ECOG (Eastern Cooperative Oncology Group) performance status of </= 1.
* Adequate renal function defined as GFR (Glomerular Filtration Rate) >/= 50 mL/min.
* Use of adequate contraception
* ECG (Electrocardiogram) within normal limits.
* Subjects must agree not to take any new vitamin supplements or herbal remedy during the study period.
* Subjects must be able to safety take lithium carbonate for at least 4 weeks before scheduled prostatectomy.

Exclusion Criteria:

* Subjects who have received any investigational medication within 30 days of first lithium dose.
* Subjects currently receiving, or who have had previous hormonal, chemotherapy or radiotherapy for prostate cancer.
* Subjects with known brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lithium carbonate.
* Uncontrolled intercurrent illness such as ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Observe any change to Performance Status and Adverse Events related to Lithium | Weekly for 4 weeks prior to radical prostatectomy and continuing for 1 - 2 weeks after surgery
  To determine the safety and tolerability of lithium in subjects with clinically localized prostate cancer.

SECONDARY OUTCOMES:
Serum lithium levels | Weekly for up to 4 weeks prior to radical prostatectomy
  To document observed levels of lithium in the serum

OTHER OUTCOMES:
Tumor response by lithium concentration | Sample collected during surgery and up to 4 weeks after baseline
  To evaluate tumor response by lithium concentration in the surgically removed prostate and serum PSA levels.

CONTACTS AND LOCATIONS:
Overall Officials: Moben Mirza, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States